CLINICAL TRIAL: NCT00567151
Title: Detection of Nontuberculous Mycobacterial co-Infection Using Duplex PCR for Mycobacterial Hsp 65 Gene and Its Clinical Significance in Patients With Smear Positive Pulmonary Tuberculosis
Brief Title: Co-Infection of NTM in Patients With Smear Positive Pulmonary TB
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Jae-Joon Yim/Associate Professor, Division of Pulmonary and Critical Care Medicine, Seoul National University Hospital
Other Study IDs: H-0711-022-225; Non-applicable
Record Dates: First submitted 2007-12-02; First posted 2007-12-04 (Estimated); Last update posted 2009-06-23 (Estimated); Status verified 2009-06

CONDITIONS: Tuberculosis, Pulmonary
MeSH Terms: conditions — Tuberculosis, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Sputa with positive AFB smear
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to elucidate the prevalence of nontuberculous mycobacterial (NTM) co-infection in patients with smear positive pulmonary TB. To detect the NTM co-infection, we will perform duplex PCR targeted for mycobacterial hsp 65 gene using sputa. In addition, the clinical significance of this co-infection will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* New patients with pulmonary TB
* Sputum AFB smear-positivity

Exclusion Criteria:

* Non-applicable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients visited Seoul National University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2007-12; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Joon Yim, MD, Principal Investigator — Seoul National Univeristy Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea